CLINICAL TRIAL: NCT02619903
Title: The Oral Microbiota as Reservoir for Systemic Opportunistic Pathogens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Daniel Joensson, Assistant professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-279
Record Dates: First submitted 2015-11-29; First posted 2015-12-02 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: COPD Exacerbation; Pulmonary Disease, Chronic Obstructive; Dental Plaque
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Test versus control for dental treatment in attenuating exacerbations in COPD.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD Control (No Intervention): Subjects with COPD recieve no treatment. When exiting the trial after 12 months, they do however receive the intervention.
- COPD Test (Active Comparator): Subjects with COPD that do get the additional dental cleaning, as well as dental examination.
  Interventions: Procedure: Dental cleaning

INTERVENTIONS:
Procedure: Dental cleaning — Dental scaling and cleaning to remove dental plaque as well as removing the tongue biofilm.
  Arms: COPD Test

SUMMARY:
Small pilot studies with approximately 20 people per group support that eradication of the oral flora causes fewer exacerbations in chronic obstructive pulmonary disease (COPD) patients. The biological underpinning put forward is that eradicating the oral microbiome will eliminate a source of re-infection as the concentration of antibiotics prescribed to treat COPD exacerbations are not able to inhibit the bacteria in the oral biofilms that require 250 times higher concentration.

The specific aim is to investigate if adding advanced dental cleaning to COPD treatment can (i) lower the number of exacerbations and (ii) improve the COPD symptoms the coming 12 months. In an effort to explain the underpinning mechanism we will collect oral dental biofilm samples at baseline and follow up in the treatment and control group to investigate changes in the composition of the biofilm.

The subjects are selected by experienced COPD nurses. Exclusion criteria are having metastatic cancer or dementia. The COPD clinic informs the dental personal about COPD parameters, including spirometry data. At the dental clinic the patient answers a questionnaire, including a COPD assessment test (CAT) which has been validated extensively. The patients undergo a dental examination and are then randomized to test or control group. The test group go through supra- and subgingival scaling and scraping of the tongue as well as chlorhexidine rinse. The control group attends all visits.

All subjects go through the intervention after 6 months and are followed up after 12 and 24 months using questionnaire, dental plaque sampling and spirometry. The COPD nurses reviewing their medical records assess number of exacerbations.

A confirmation of the study hypothesis will be important in lowering the number of exacerbations in COPD patients, causing less suffering, less costs and less usage of antibiotics. If dental treatment is beneficial for exacerbation frequency it could be argued that dental treatment should be subsidized in this patient category.

DETAILED DESCRIPTION:
Introduction The dental biofilm offers a protected environment for bacteria during systemic antibiotic treatment and may consequently be a source of reinfection. The concentration of antibiotic needed for inhibiting the growth of bacteria within a dental biofilm has been estimated to be 250 times greater than for planktonically growing bacteria (1). Chronic obstructive pulmonary disease (COPD) exacerbations cause pain and discomfort for the patient, healthcare resources and an increased usage of antibiotics. Smaller studies indicate that the act of advanced dental cleaning may lower the risk of reinfected COPD, but this needs to be validated in a larger randomized study to promote clinical implications.

COPD is a growing health problem worldwide. In 2020, COPD is projected to rank fifth in terms of burden of disease and third in terms of mortality (2). Assessment of COPD is based on the patient´s level of symptoms, exacerbation history and severity of spirometric abnormality. In a randomly selected Swedish cohort, the prevalence of COPD was 16.2%, and 34% of the COPD patients had never smoked (3). Unfortunately, none of the existing medications for COPD has been shown conclusively to modify the long-term decline in lung-function, but COPD patients are usually prescribed β2-adrenerg receptor agonists and anticholinergics (2). For acute exacerbations, the patients have oral steroids and antibiotics, typically doxycycline and amoxicillin. Importantly, two smaller (n=20 per group) pilot studies (4,5) have reported a lower frequency of exacerbations in COPD patients that have received advanced dental cleaning, suggesting that the oral microbiome might constitute a reservoir that infects the lungs in COPD. There is a need of studies based on larger cohorts in order to claim that dental treatment should be added to the treatment regime of COPD, to decrease the frequencies of exacerbations and thereby minimize physical suffering as well as related costs.

Hypothesis The hypothesis of this project is that adding advanced dental cleaning to established COPD treatment regime delays and lowers the frequency of exacerbations by eliminating a source of reinfections.

Aim The overall aim of this project is to investigate if the treatment of COPD can be optimized by adding advanced dental cleaning to the established treatment regime and thereby eliminate a source of reinfections.

The specific aim is to investigate if adding advanced dental cleaning to COPD treatment can (i) lower the number of exacerbations and (ii) improve the COPD symptoms the coming 6 and 12 months. In an effort to explain the underpinning mechanism we will collect oral dental biofilm samples at baseline and follow up in the treatment and control group to investigate changes in the composition of the biofilm.

COPD project At the lung clinic The COPD project will be conducted at Region Skane lung clinic and in collaboration with the COPD clinics in Skne In Örebro the subjects will be recruited from the lung clinic in collaboration with Dr. Josefin Sundh and the dental cleaning will be performed at the dental specialist clinic, folktandvarden Örebro. A COPD patient will be informed about the current study by a nurse. The patient will be asked to sign a consent and handed the written information including the number to the dental clinic.

At the dental clinic The dental clinic receives a phone call from the person who just signed a consent; alternatively, a nurse at the dental clinic calls the patient. At the dental clinic the patient is randomized to, either the advanced dental cleaning group, or a control group by the dentist or dental hygienist at the dental clinic. When the patient comes to the dental visit, both groups undergo a periodontal examination and microbiological sampling.

Questionnaire - Upon arriving at the dental clinic, the participant is asked to fill out a questionnaire that includes medical history and CAT-questionnaire.

The microbiological sampling is done by collecting the GenoTek tube by sampling the dental plaque samples.

Periodontal examination is performed on 6 sites per tooth including the third molar. Periodontal pockets ≥ 4mm are registered as well as bleeding upon probing, plaque index and attachment loss.

Intervention - The oral biofilm will be disrupted and removed on the sub- as well as supragingival surfaces of the teeth. Supragingival surfaces will be cleaned using the prophylactic paste RDA 250 supplemented with curettes and ultrasonic debridement. Subgingival surfaces will be cleaned using curettes and ultrasonic debridement when indicated based on the periodontal examination. The tongue will be cleaned using a tongue scraper. Finally, the patient will be asked to rinse 10 ml of 2 mg/ml chlorhexidine mouth rinse for one minute.

Follow-up - After 6 months, 12 months and 24 months the participants revisits the dental clinic. They fill out a new CAT form and a questionnaire asking how many exacerbations that needed medical attention since they joined the study (this is double checked in their medical records), if they have taken antibiotics for any other reason or changed their medications in any way. They are also asked about any dental treatments.

Microbiological analysis The subsequent microbiological analysis will be executed using deep sequencing, as well as qPCR.

Time schedule 2016-2017 - Participants are recruited, randomized and the treatment group is treated. 2017-2020 - Participants are followed up.

2020 - Data analysis and publication.

Network Daniel Jönsson - PhD in 2007 and a postdoc on the systemic effects of periodontal disease in 2009 and 2010 at Columbia University, New York, NY, USA. Became a specialist in periodontics in 2014 and currently positioned at Malmö University and Region Skane, Lund. Dr. Jönsson will start a part time position in Örebro in 2016.

Bodil Ohlsson - Professor and specialist in Internal Medicine and Gastroenterology at Lund University and Region Skane University hospital.

Hanan Tanash - PhD and specialist in Internal Medicine. Field of interest - COPD.

Josefin Sundh - Associate Professor at Örebro University hospital. Field of interest - COPD.

Frida Fak - Associate Professor at Lund University. Field of interest - microbiology.

Folktandvarden Skane - two dental hygienists have been recruited for the project.

Folktandvarden Örebro - a post-graduate student is being recruited for the dental cleaning as well as managing the logistics of the project. Daniel Jönsson will be the supervisor of the student.

Power analysis In a power analysis based on the standard deviations from the pilot study of Kucukoskun et al. [3] indicated 80% power to detect a difference of p<0.05 of 1.5 exacerbations per year in a sample of 49 subjects in each group.

Significance As antibiotics is part of the COPD treatment regime this study may restrict the usage of antibiotics, minimizing antibiotic resistance. COPD exacerbations disable the person to go to work which causes financial consequences, but also healthcare expenses. Most importantly, the study will plausibly improve life quality and extend the life span of patients suffering from COPD. We already have preliminary data that subjects in the treatment group have an OR 3.9 for being stable or having less COPD-symptoms in this progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* COPD arm - COPD Gold standard 1-4.

Exclusion Criteria:

* Physically unable to make it to the dental clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-02; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
COPD exacerbations in 12 months | 12 months
  We will ask the patients how many exacerbations they had and go through medical records.

SECONDARY OUTCOMES:
COPD symptoms | 12 months
  COPD symptoms based on CAT-score (COPD Assessment Test)

OTHER OUTCOMES:
Changes in oral microbiome | 12 months
  Changes in the oral plaque microbiota comparing baseline and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jönsson, DDS, PhD, Principal Investigator — Lund University
Locations (2):
- Sweden (2):
  - Folktandvarden Skane, Malmo
  - Orebro Specialisttandvard, Örebro

IPD SHARING:
Plan to Share IPD: No